CLINICAL TRIAL: NCT00925015
Title: A Phase I Study of MK-0646 in Combination With Cetuximab and Irinotecan in Patients With Advanced or Metastatic Colorectal Cancer
Brief Title: Phase I Study of Dalotuzumab (MK-0646) in Combination With Cetuximab and Irinotecan in Participants With Colorectal Cancer (MK-0646-016)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0646-016; 2009_602
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — dalotuzumab; Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cetux/Irin - Dmab 10 mg/kg (Experimental): After treatment with Cetuximab (Cetux) and Irinotecan (Irin), Dalotuzumab (Dmab) was administered as an intravenous infusion at 10 mg/kg in Cycle 1 on Days 22, 29 and 36; followed in subsequent cycles by treatment with 10 mg/kg on Days 1, 8, 15, 22, 29 and 36. Each cycle was 6 weeks long.
  Interventions: Biological: Dalotuzumab 10 mg/kg; Biological: Cetuximab; Drug: Irinotecan
- Cetux/Irin - Dmab 15/7.5 mg/kg (Experimental): After treatment with Cetux/Irin, Dmab was administered as an intravenous infusion at 15 mg/kg in Cycle 1 on Days 8, 22 and 36; followed in subsequent cycles by treatment with 7.5 mg/kg on Days 8, 22 and 36. Each cycle was 6 weeks long.
  Interventions: Biological: Cetuximab; Drug: Irinotecan; Biological: Dalotuzumab 15/7.5 mg/kg
- Dmab 10 mg/kg - Cetux/Irin (DDI) (Experimental): Dmab was administered in each cycle as an intravenous infusion at 10 mg/kg once weekly on Days 1, 22 and 29; followed by treatment with Cetux/Irin. For Drug-Drug Interaction (DDI). Each cycle was 6 weeks long.
  Interventions: Biological: Dalotuzumab 10 mg/kg; Biological: Cetuximab; Drug: Irinotecan

INTERVENTIONS:
Biological: Dalotuzumab 10 mg/kg — Dalotuzumab at 10 mg/kg was intravenously administered once weekly
  Other Names: MK-0646
  Arms: Cetux/Irin - Dmab 10 mg/kg; Dmab 10 mg/kg - Cetux/Irin (DDI)
Biological: Cetuximab — Following pre-treatment with a histamine-receptor antagonist, Cetuximab was administered with an initial intravenous infusion of 400 mg/m^2, followed by subsequent once weekly intravenous infusions of 250 mg/m^2
Drug: Irinotecan — Irinotecan was administered with an intravenous infusion of 150 mg/m^2, once every other week for 42 days
Biological: Dalotuzumab 15/7.5 mg/kg — Dalotuzumab was intravenously administered, with the first infusion of 15 mg/kg, followed by subsequent infusions of 7.5 mg/kg
  Other Names: MK-0646
  Arms: Cetux/Irin - Dmab 15/7.5 mg/kg

SUMMARY:
The purposes of this study were to assess the safety, tolerability, pharmacokinetic interactions, and the Human Anti-Human Antibody of dalotuzumab in combination with cetuximab and irinotecan in participants with advanced or metastatic colorectal cancer in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Is 20 years of Age or older
* Has a histologically or cytologically confirmed colorectal cancer
* Has previously failed both Irinotecan and Oxaliplatin containing regimens and should have progressed on or within 3 months of completing their last line of therapy with objective radiological evidence of progression as verified by previous radiologic scans
* Must have adequate organ function

Exclusion Criteria:

* Has had chemotherapy, radiotherapy, or biological therapy within 4 weeks prior to initial dosing on this study or whose toxicities from agents administrated 4 weeks earlier have not resolved to at least grade 1 or baseline
* Has experienced intolerable toxicity to Irinotecan therapy
* Has prior exposure to insulin-like growth factor 1 receptor (IGF-1R) inhibitors or epidermal growth factor receptor (EGFR) inhibitors (e.g. Cetuximab)
* Is concurrently using growth hormone (GH), Or GH inhibitors

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06-17 (Actual); Primary Completion 2010-07-28 (Actual); Study Completion 2010-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Doi T, Muro K, Yoshino T, Fuse N, Ura T, Takahari D, Feng HP, Shimamoto T, Noguchi K, Ohtsu A. Phase 1 pharmacokinetic study of MK-0646 (dalotuzumab), an anti-insulin-like growth factor-1 receptor monoclonal antibody, in combination with cetuximab and irinotecan in Japanese patients with advanced colorectal cancer. Cancer Chemother Pharmacol. 2013 Sep;72(3):643-52. doi: 10.1007/s00280-013-2240-8. Epub 2013 Aug 7. PMID 23921573

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetux/Irin - Dmab 15/7.5 mg/kg: After treatment with Cetux/Irin, Dmab was administered as an intravenous infusion at 15 mg/kg in Cycle 1 on Day 8; followed in subsequent infusions by treatment with 7.5 mg/kg on Days 22 and 36. Each cycle was 6 weeks long.
- Dmab 10 mg/kg - Cetux/Irin (DDI): Dmab was administered in each cycle as an intravenous infusion at 10 mg/kg once weekly on Days 1, 22 and 29; followed by treatment with Cetux/Irin. Each cycle was 6 weeks long. For Drug-Drug Interaction (DDI).
Period: Overall Study
Arm/Group | Cetux/Irin - Dmab 10 mg/kg | Cetux/Irin - Dmab 15/7.5 mg/kg | Dmab 10 mg/kg - Cetux/Irin (DDI)
Started | 8 | 6 | 6
Completed | 0 | 0 | 0
Not Completed | 8 | 6 | 6
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Progressive Disease | 7 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetux/Irin - Dmab 10 mg/kg | Cetux/Irin - Dmab 15/7.5 mg/kg | Dmab 10 mg/kg - Cetux/Irin (DDI) | Total
Number analyzed (Participants) | 8 | 6 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (5.6) | 59.3 (3.6) | 59.7 (8.5) | 60.6 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 5
  Male | 5 | 5 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose-limiting Toxicities (DLTs)
Description: To be declared a DLT an adverse experience had a causality related to study therapy. DLTs could be adverse experiences possibly, probably, or definitely related to study therapy by the Investigator, and included the following : Grade 4 neutropenia lasting >= 5 days; Grade 3 or 4 neutropenia with fever >38.5°C; Grade 4 thrombocytopenia; Grade 3 or Grade 4 non-hematologic toxicity, except inadequately treated diarrhea, nausea and vomiting, rash, hyperglycemia, and transient abnormality of electrolytes. Anemia, infusion reactions, hypersensitivity reactions, and adverse experiences not-related to study therapy did not qualify as DLTs.
Time Frame: Four weeks of Cycle 1 treatment (up to 28 days)
Population: Participants treated with study medication. The Dmab 10 mg/kg - Cetux/Irin arm was not evaluated. In the Cetux/Irin - Dmab 10 mg/kg (DDI) arm two participants were not analyzed because one had febrile neutropenia (Grade 3) before the first treatment, and the second had a skin toxicity (Grade 3) before the DLT evaluation period.
Measure: Number; unit: DLT
Groups:
- Cetux/Irin - Dmab 10 mg/kg: After treatment with Cetuximab (Cetux) and Irinotecan (Irin), Dalotuzumab (Dmab) was administered as an intravenous infusion at 10 mg/kg in cycle 1 on Days 22, 29 and 36; followed in subsequent cycles by treatment with 10 mg/kg on Days 1,8, 15, 22, 29 and 36.
- Dmab 10 mg/kg - Cetux/Irin (DDI): Dmab was administered in each cycle as an intravenous infusion at 10 mg/kg once weekly on Days 1, 22 and 29; followed by treatment with Cetux/Irin. For DDI.
Arm/Group | Cetux/Irin - Dmab 10 mg/kg | Cetux/Irin - Dmab 15/7.5 mg/kg | Dmab 10 mg/kg - Cetux/Irin (DDI)
Number analyzed (Participants) | 6 | 6 | 0
DLT | 0 | 1 |

2. Secondary Outcome: Number of Participants With Human Anti-Human Antibody (HAHA)
Description: Sera were collected from participants prior to administration of the first dose of study drug, every 6 weeks during the study period, then 4 weeks, 8 weeks and 12 weeks post-treatment. A sandwich format enzyme-linked immunosorbent assay (ELISA) was used to detect the presence of HAHA in serum.
Time Frame: Up to 12 weeks after the last administration of dalotuzumab (up to 349 days)
Population: All treated participants, excluding those without measurable data.
Measure: Number; unit: Participants
Arm/Group | Cetux/Irin - Dmab 10 mg/kg | Cetux/Irin - Dmab 15/7.5 mg/kg | Dmab 10 mg/kg - Cetux/Irin (DDI)
Number analyzed (Participants) | 8 | 6 | 6
Participants | 0 | 0 | 0

3. Secondary Outcome: Time to Maximum Concentration (Tmax) of Dalotuzumab Following Administration of 10 mg/kg Dalotuzumab Alone in or in Combination With Cetuximab / Irinotecan
Description: In Cycle 1 Dalotuzumab was administered on Days 1 and 22 as an intravenous infusion at 10 mg/kg. In the same Cycle 1 Cetuximab was administered on Days 8, 15, 22 and 29; and Irinotecan was administered on Days 8 and 22. The Tmax of plasma Dalotuzumab alone was determined on Day 1, and in combination with cetuximab/irinotecan on Day 22.
Time Frame: Cycle 1: Day 1 and Day 22 at predose, 0.5 h after start of infusion, end of infusion, 5, 8, 24, 30, 48, 96 and 168 h after initiation of dalotuzumab infusion
Population: Participants from the Dmab 10 mg/kg - Cetux/Irin (DDI) arm only, who were treated with study medication and had evaluable measurements at baseline and at least once during treatment. No explicit imputation was made for missing data.
Measure: Median (Full Range); unit: h
Groups:
- Dalotuzumab 10 mg/kg Alone: Participants were treated in Cycle 1, Day 1 with Dalotuzumab alone
- Dalotuzumab 10 mg/kg + Cetuximab/Irinotecan: Participants were treated in Cycle 1, Day 22 with both Dalotuzumab + Cetuximab/Irinotecan
Arm/Group | Dalotuzumab 10 mg/kg Alone | Dalotuzumab 10 mg/kg + Cetuximab/Irinotecan
Number analyzed (Participants) | 6 | 6
h | 5.0 [2.0 to 8.0] | 3.5 [2.0 to 24.0]

4. Secondary Outcome: Concentration at the End of Infusion (Ceoi) of Dalotuzumab Following Administration of 10 mg/kg Dalotuzumab Alone or in Combination With Cetuximab / Irinotecan
Description: In Cycle 1 Dalotuzumab was administered on Days 1 and 22 as an intravenous infusion at 10 mg/kg. In the same Cycle 1 Cetuximab was administered on Days 8, 15, 22 and 29; and Irinotecan was administered on Days 8 and 22. The Ceoi of plasma Dalotuzumab alone was determined on Day 1, and in combination with cetuximab/irinotecan on Day 22.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Dalotuzumab 10 mg/kg Alone | Dalotuzumab 10 mg/kg + Cetuximab/Irinotecan
Number analyzed (Participants) | 6 | 6
µg/mL | 211.2 (14.3) [2.0 to 8.0] | 267.3 (27.1) [2.0 to 24.0]

5. Secondary Outcome: Maximum Concentration (Cmax) of Dalotuzumab Following Administration of 10 mg/kg Dalotuzumab Alone or in Combination With Cetuximab / Irinotecan
Description: In Cycle 1 Dalotuzumab was administered on Days 1 and 22 as an intravenous infusion at 10 mg/kg. In the same Cycle 1 Cetuximab was administered on Days 8, 15, 22 and 29; and Irinotecan was administered on Days 8 and 22. The Cmax of plasma Dalotuzumab alone was determined on Day 1, and in combination with cetuximab/irinotecan on Day 22.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Dalotuzumab 10 mg/kg Alone | Dalotuzumab 10 mg/kg + Cetuximab/Irinotecan
Number analyzed (Participants) | 6 | 6
µg/mL | 247.6 (14.4) [2.0 to 8.0] | 311.9 (21.3) [2.0 to 24.0]

6. Secondary Outcome: Apparent Terminal Half-life (T1/2) of Dalotuzumab Following Administration of 10 mg/kg Dalotuzumab Alone or in Combination With Cetuximab / Irinotecan
Description: In Cycle 1 Dalotuzumab was administered on Days 1 and 22 as an intravenous infusion at 10 mg/kg. In the same Cycle 1 Cetuximab was administered on Days 8, 15, 22 and 29; and Irinotecan was administered on Days 8 and 22. The T1/2 of plasma Dalotuzumab alone was determined on Day 1, and in combination with cetuximab/irinotecan on Day 22.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Dalotuzumab 10 mg/kg Alone | Dalotuzumab 10 mg/kg + Cetuximab/Irinotecan
Number analyzed (Participants) | 6 | 6
h | 131.4 (21.5) [2.0 to 8.0] | 141.4 (32.1) [2.0 to 24.0]

7. Secondary Outcome: Clearance From Plasma (CL) of Dalotuzumab Following Administration of 10 mg/kg Dalotuzumab Alone or in Combination With Cetuximab / Irinotecan
Description: In Cycle 1 Dalotuzumab was administered on Days 1 and 22 as an intravenous infusion at 10 mg/kg. In the same Cycle 1 Cetuximab was administered on Days 8, 15, 22 and 29; and Irinotecan was administered on Days 8 and 22. The CL of plasma Dalotuzumab alone was determined on Day 1, and in combination with cetuximab/irinotecan on Day 22.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min/kg
Arm/Group | Dalotuzumab 10 mg/kg Alone | Dalotuzumab 10 mg/kg + Cetuximab/Irinotecan
Number analyzed (Participants) | 6 | 6
mL/min/kg | 0.0049 (21.9) [2.0 to 8.0] | 0.0038 (33.7) [2.0 to 24.0]

8. Secondary Outcome: Steady-state Volume of Distribution (Vss) of Dalotuzumab Following Administration of 10 mg/kg Dalotuzumab Alone or in Combination With Cetuximab / Irinotecan
Description: In Cycle 1 Dalotuzumab was administered on Days 1 and 22 as an intravenous infusion at 10 mg/kg. In the same Cycle 1 Cetuximab was administered on Days 8, 15, 22 and 29; and Irinotecan was administered on Days 8 and 22. The Vss of plasma Dalotuzumab alone was determined on Day 1, and in combination with cetuximab/irinotecan on Day 22.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | Dalotuzumab 10 mg/kg Alone | Dalotuzumab 10 mg/kg + Cetuximab/Irinotecan
Number analyzed (Participants) | 6 | 6
L/kg | 0.0558 (11.1) [2.0 to 8.0] | 0.0459 (14.2) [2.0 to 24.0]

9. Secondary Outcome: Area Under the Concentration-time Curve From 0-24 Hours Post-dose (AUC0-24) of Dalotuzumab Following Administration of 10 mg/kg Dalotuzumab Alone or in Combination With Cetuximab / Irinotecan
Description: In Cycle 1 Dalotuzumab was administered on Days 1 and 22 as an intravenous infusion at 10 mg/kg. In the same Cycle 1 Cetuximab was administered on Days 8, 15, 22 and 29; and Irinotecan was administered on Days 8 and 22. The AUC0-24 of plasma Dalotuzumab alone was determined on Day 1, and in combination with cetuximab/irinotecan on Day 22.
Time Frame: Cycle 1: Day 1 and Day 22 at predose, 0.5 h after start of infusion, end of infusion, 5, 8 and 24 h after initiation of dalotuzumab infusion
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/mL
Arm/Group | Dalotuzumab 10 mg/kg Alone | Dalotuzumab 10 mg/kg + Cetuximab/Irinotecan
Number analyzed (Participants) | 6 | 6
mg*h/mL | 4.56 (11.7) [2.0 to 8.0] | 5.39 (18.8) [2.0 to 24.0]

10. Secondary Outcome: Area Under the Concentration-time Curve From 0-168 Hours Post-dose (AUC0-168) of Dalotuzumab Following Administration of 10 mg/kg Dalotuzumab Alone or in Combination With Cetuximab / Irinotecan
Description: In Cycle 1 Dalotuzumab was administered on Days 1 and 22 as an intravenous infusion at 10 mg/kg. In the same Cycle 1 Cetuximab was administered on Days 8, 15, 22 and 29; and Irinotecan was administered on Days 8 and 22. The AUC0-168 of plasma Dalotuzumab alone was determined on Day 1, and in combination with cetuximab/irinotecan on Day 22.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/mL
Arm/Group | Dalotuzumab 10 mg/kg Alone | Dalotuzumab 10 mg/kg + Cetuximab/Irinotecan
Number analyzed (Participants) | 6 | 6
mg*h/mL | 19.6 (13.1) [2.0 to 8.0] | 24.5 (19.0) [2.0 to 24.0]

11. Secondary Outcome: Tmax of Cetuximab Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Cetuximab was administered with an initial intravenous infusion of 400 mg/m^2 on Day 8, followed by subsequent once weekly intravenous infusions of 250 mg/m^2 on Days 15, 22, 29 and 36. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Irinotecan was administered on Days 1, 22, and 29. The Tmax of plasma Cetuximab was determined alone on Day 15 and in combination with dalotuzumab on Day 29.
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 2, 5, 8, 24, 48, 96 and 168 h after initiation of cetuximab infusion
Population: Participants from the Cetux/Irin - Dmab 10 mg/kg arm only, who were treated with study medication and had evaluable measurements at baseline and at least once during treatment. No explicit imputation was made for missing data.
Measure: Median (Full Range); unit: h
Groups:
- Cetuximab/Irinotecan Alone: Participants were treated in Cycle 1, Day 15 with Cetuximab/Irinotecan alone
- Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg: Participants previously treated with Cetuximab/Irinotecan were treated in Cycle 1, Day 29 with Dalotuzumab 10 mg/kg
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
h | 7.9 [2.0 to 8.0] | 2.0 [2.0 to 2.1]

12. Secondary Outcome: Cmax of Cetuximab Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Cetuximab was administered with an initial intravenous infusion of 400 mg/m^2 on Day 8, followed by subsequent once weekly intravenous infusions of 250 mg/m^2 on Days 15, 22, 29 and 36. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Irinotecan was administered on Days 1, 22, and 29. The Cmax of plasma Cetuximab was determined alone on Day 15 and in combination with dalotuzumab on Day 29.
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 2, 5, 8, 24, 48, 96 and 168 h after initiation of cetuximab infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
µg/mL | 204.0 (15.0) [2.0 to 8.0] | 236.5 (23.0) [2.0 to 2.1]

13. Secondary Outcome: T1/2 of Cetuximab Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Cetuximab was administered with an initial intravenous infusion of 400 mg/m^2 on Day 8, followed by subsequent once weekly intravenous infusions of 250 mg/m^2 on Days 15, 22, 29 and 36. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Irinotecan was administered on Days 1, 22, and 29. The T1/2 of plasma Cetuximab was determined alone on Day 15 and in combination with dalotuzumab on Day 29.
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 2, 5, 8, 24, 48, 96 and 168 h after initiation of cetuximab infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
h | 129.4 (26.0) [2.0 to 8.0] | 131.9 (34.5) [2.0 to 2.1]

14. Secondary Outcome: CL of Cetuximab Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Cetuximab was administered with an initial intravenous infusion of 400 mg/m^2 on Day 8, followed by subsequent once weekly intravenous infusions of 250 mg/m^2 on Days 15, 22, 29 and 36. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Irinotecan was administered on Days 1, 22, and 29. The CL of plasma Cetuximab was determined alone on Day 15 and in combination with dalotuzumab on Day 29.
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 2, 5, 8, 24, 48, 96 and 168 h after initiation of cetuximab infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/m^2
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
mL/h/m^2 | 7.81 (32.8) [2.0 to 8.0] | 6.82 (40.5) [2.0 to 2.1]

15. Secondary Outcome: Vss of Cetuximab Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Cetuximab was administered with an initial intravenous infusion of 400 mg/m^2 on Day 8, followed by subsequent once weekly intravenous infusions of 250 mg/m^2 on Days 15, 22, 29 and 36. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Irinotecan was administered on Days 1, 22, and 29. The Vss of plasma Cetuximab was determined alone on Day 15 and in combination with dalotuzumab on Day 29.
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 2, 5, 8, 24, 48, 96 and 168 h after initiation of cetuximab infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/m^2
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
L/m^2 | 1.45 (10.0) [2.0 to 8.0] | 1.32 (17.8) [2.0 to 2.1]

16. Secondary Outcome: AUC0-24 of Cetuximab Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Cetuximab was administered with an initial intravenous infusion of 400 mg/m^2 on Day 8, followed by subsequent once weekly intravenous infusions of 250 mg/m^2 on Days 15, 22, 29 and 36. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Irinotecan was administered on Days 1, 22, and 29. The AUC0-24 of plasma Cetuximab was determined alone on Day 15 and in combination with dalotuzumab on Day 29.
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 2, 5, 8 and 24 h after initiation of cetuximab infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/mL
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
mg*h/mL | 4.02 (14.5) [2.0 to 8.0] | 4.12 (26.1) [2.0 to 2.1]

17. Secondary Outcome: AUC0-168 of Cetuximab Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Cetuximab was administered with an initial intravenous infusion of 400 mg/m^2 on Day 8, followed by subsequent once weekly intravenous infusions of 250 mg/m^2 on Days 15, 22, 29 and 36. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Irinotecan was administered on Days 1, 22, and 29. The AUC0-168 of plasma Cetuximab was determined alone on Day 15 and in combination with dalotuzumab on Day 29.
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 2, 5, 8, 24, 48, 96 and 168 h after initiation of cetuximab infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/mL
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
mg*h/mL | 18.6 (20.9) [2.0 to 8.0] | 20.1 (28.6) [2.0 to 2.1]

18. Secondary Outcome: Tmax of Irinotecan Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Irinotecan was administered with an intravenous infusion of 150 mg/m^2 once every other week on Days 1, 15, and 29. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Cetuximab was administered on Days 1, 8, 15, 22, 29 and 36. The Tmax of plasma Irinotecan was determined alone on Day 15 and in combination with dalotuzumab on Day 29.
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 1, 5, 8, 24, and 48 h after completion of Irinotecan infusion
Population: as for outcome 11
Measure: Median (Full Range); unit: h
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
h | 1.0 [0.97 to 1.0] | 1.0 [1.0 to 1.1]

19. Secondary Outcome: Cmax of Irinotecan Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Irinotecan was administered with an intravenous infusion of 150 mg/m^2 once every other week on Days 1, 15, and 29. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Cetuximab was administered on Days 1, 8, 15, 22, 29 and 36. The Cmax of plasma Irinotecan was determined alone on Day 15 and in combination with dalotuzumab on Day 29.
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 1, 5, 8, 24, and 48 h after completion of Irinotecan infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
µg/mL | 1.21 (22.8) [0.97 to 1.0] | 1.13 (25.6) [1.0 to 1.1]

20. Secondary Outcome: T1/2 of Irinotecan Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Irinotecan was administered with an intravenous infusion of 150 mg/m^2 once every other week on Days 1, 15, and 29. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Cetuximab was administered on Days 1, 8, 15, 22, 29 and 36. The T1/2 of plasma Irinotecan was determined alone on Day 15 and in combination with dalotuzumab on Day 29..
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 1, 5, 8, 24, and 48 h after completion of Irinotecan infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
h | 8.95 (9.13) [0.97 to 1.0] | 9.67 (12.7) [1.0 to 1.1]

21. Secondary Outcome: CL of Irinotecan Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Irinotecan was administered with an intravenous infusion of 150 mg/m^2 once every other week on Days 1, 15, and 29. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Cetuximab was administered on Days 1, 8, 15, 22, 29 and 36. The CL of plasma Irinotecan was determined alone on Day 15 and in combination with dalotuzumab on Day 29.
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 1, 5, 8, 24, and 48 h after completion of Irinotecan infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/m^2
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
L/h/m^2 | 12.3 (35.7) [0.97 to 1.0] | 13.1 (34.3) [1.0 to 1.1]

22. Secondary Outcome: Vss of Irinotecan Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Irinotecan was administered with an intravenous infusion of 150 mg/m^2 once every other week on Days 1, 15, and 29. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Cetuximab was administered on Days 1, 8, 15, 22, 29 and 36. The Vss of plasma Irinotecan was determined alone on Day 15 and in combination with dalotuzumab on Day 29.
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 1, 5, 8, 24, and 48 h after completion of Irinotecan infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/m^2
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
L/m^2 | 117 (27.5) [0.97 to 1.0] | 137 (24.9) [1.0 to 1.1]

23. Secondary Outcome: AUC0-24 of Irinotecan Following Administration of Cetuximab / Irinotecan Alone, or in Combination With 10 mg/kg Dalotuzumab
Description: In Cycle 1 Irinotecan was administered with an intravenous infusion of 150 mg/m^2 once every other week on Days 1, 15, and 29. In the same Cycle 1 Dalotuzumab 10 mg/kg was administered on Days 22, 29 and 36; and Cetuximab was administered on Days 1, 8, 15, 22, 29 and 36. The AUC0-24 of plasma Irinotecan was determined alone on Day 15 and in combination with dalotuzumab on Day 29.
Time Frame: Cycle 1: Day 15 and Day 29 at predose, 1, 5, 8 and 24 h after completion of Irinotecan infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cetuximab/Irinotecan Alone | Cetuximab/Irinotecan + Dalotuzumab 10 mg/kg
Number analyzed (Participants) | 7 | 6
µg*h/mL | 7.19 (33.6) [0.97 to 1.0] | 6.64 (31.9) [1.0 to 1.1]

24. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product, is also an AE.
Time Frame: Approximately 4 weeks after last drug treatment (up to Day 293)
Population: Participants treated with study medication.
Measure: Number; unit: Participants
Arm/Group | Cetux/Irin - Dmab 10 mg/kg | Cetux/Irin - Dmab 15/7.5 mg/kg | Dmab 10 mg/kg - Cetux/Irin (DDI)
Number analyzed (Participants) | 8 | 6 | 6
Participants | 8 | 6 | 6

ADVERSE EVENTS:
Time Frame: Approximately 4 weeks after last drug treatment (up to Day 293)
Description: Participants treated with one or more doses of study medication.
Groups:
- Cetux/Irin - Dalotuzumab 10 mg/Kg: After treatment with Cetux and Irin, Dmab was administered as an intravenous infusion at 10 mg/kg in Cycle 1 on Days 22, 29 and 36; followed in subsequent cycles by treatment with 10 mg/kg on Days 1, 8, 15, 22, 29 and 36. Each cycle was 6 weeks long.
- Cetux/Irin - Dalotuzumab 15/7.5 mg/Kg: After treatment with Cetux/Irin, Dmab was administered as an intravenous infusion at 15 mg/kg in Cycle 1 on Days 8, 22 and 36; followed in subsequent cycles by treatment with 7.5 mg/kg on Days 8, 22 and 36. Each cycle was 6 weeks long.
- Dalotuzumab 10 mg/Kg - Cetux/Irin (DDI): Dmab was administered in each cycle as an intravenous infusion at 10 mg/kg once weekly on Days 1, 22 and 29; followed by treatment with Cetux/Irin. Each cycle was 6 weeks long.
Arm/Group | Cetux/Irin - Dalotuzumab 10 mg/Kg | Cetux/Irin - Dalotuzumab 15/7.5 mg/Kg | Dalotuzumab 10 mg/Kg - Cetux/Irin (DDI)
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/6 | 1/6
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetux/Irin - Dalotuzumab 10 mg/Kg (N=8) | Cetux/Irin - Dalotuzumab 15/7.5 mg/Kg (N=6) | Dalotuzumab 10 mg/Kg - Cetux/Irin (DDI) (N=6)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetux/Irin - Dalotuzumab 10 mg/Kg (N=8) | Cetux/Irin - Dalotuzumab 15/7.5 mg/Kg (N=6) | Dalotuzumab 10 mg/Kg - Cetux/Irin (DDI) (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 7 (24) | 2 (4) | 6 (18)
Lymphopenia (Blood and lymphatic system disorders) | 4 (17) | 0 (0) | 3 (6)
Neutropenia (Blood and lymphatic system disorders) | 7 (24) | 2 (4) | 5 (27)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (5) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (7) | 5 (23) | 3 (18)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (8) | 4 (8) | 3 (5)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Plicated tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 5 (7) | 3 (5) | 3 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (3) | 3 (3)
Fatigue (General disorders) | 4 (8) | 4 (9) | 2 (6)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 2 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (2) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 6 (14) | 2 (5) | 5 (16)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (9) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (7) | 0 (0) | 2 (4)
Blood alkaline phosphatase increased (Investigations) | 3 (5) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 5 (5) | 1 (1) | 2 (5)
Decreased appetite (Metabolism and nutrition disorders) | 4 (8) | 3 (9) | 2 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 3 (9) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (4) | 2 (7) | 3 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (12) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 (20) | 1 (5) | 5 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (4) | 1 (1) | 1 (3)
Skin erosion (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.